CLINICAL TRIAL: NCT00025519
Title: Submyeloablative Allogeneic Blood Stem Cell Transplantation With HLA Identical Donor Lymphocyte Infusions From Matched Related and Matched Unrelated Donors for Treatment of Metastatic Renal Cell Carcinoma
Brief Title: Peripheral Stem Cell Transplantation in Treating Patients With Metastatic or Recurrent Kidney Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: FCCC-01006; CDR0000068970 (Registry Identifier: PDQ (Physician Data Query)); TUHSC-3721; NCI-G01-2021
Record Dates: First submitted 2001-10-11; First posted 2003-01-27 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer; recurrent renal cell cancer; clear cell renal cell carcinoma
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — fludarabine phosphate; Mycophenolic Acid; Tacrolimus; Thalidomide; Peripheral Blood Stem Cell Transplantation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: therapeutic allogeneic lymphocytes
Drug: fludarabine phosphate
Drug: mycophenolate mofetil
Drug: tacrolimus
Drug: thalidomide
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Peripheral stem cell transplantation may be able to replace immune cells that were destroyed by chemotherapy and radiation therapy used to kill cancer cells. Sometimes the transplanted cells can be rejected by the body's tissues. Mycophenolate mofetil, tacrolimus, and donor white blood cells may prevent this from happening.

PURPOSE: Phase II trial to study the effectiveness of chemotherapy followed by peripheral stem cell transplantation in treating patients who have metastatic or recurrent kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of submyeloablative HLA-identical allogeneic peripheral blood stem cell transplantation in patients with metastatic or recurrent renal cell carcinoma.
* Determine the toxicity of this regimen, in terms of incidence and severity of graft rejection, acute graft-vs-host disease (GVHD), chronic GVHD, adverse effects from the preparative regimen and thalidomide, and infection and bleeding, in these patients.
* Determine the efficacy of this regimen, in terms of objective partial and complete response rates, in these patients.
* Determine the engraftment rates and extent of chimerism in patients treated with this regimen.
* Determine the overall survival and time to treatment failure rate in patients treated with this regimen.
* Determine the impact of thalidomide on the treatment of chronic GVHD in patients treated with this regimen.

OUTLINE: Patients are stratified according to risk (low vs high).

Patients receive fludarabine IV over 30 minutes once daily on days -4 to -2 followed by total body irradiation on day -1. Patients receive tacrolimus IV over 24 hours or orally daily on days -3 to 35 and oral mycophenolate mofetil twice daily on days -3 to 28 as graft-vs-host disease (GVHD) prophylaxis. Patients undergo allogeneic peripheral blood stem cell transplantation over 1-2 hours on day 0.

Patients maintaining a mixed chimerism with no evidence of grade III or IV GVHD receive donor lymphocyte infusions (DLI) on days 60, 90, and 120. Patients may receive additional DLI as needed. Patients with limited chronic GVHD receive oral thalidomide daily beginning after day 80 and continuing for 1 year or until disease progression or resolution of chronic GVHD.

Patients are followed at 1, 3, 6, and 12 months and then every 6 months thereafter.

PROJECTED ACCRUAL: A maximum of 20-40 patients (10-20 per stratum) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed renal cell carcinoma (RCC)

  * Histology demonstrates major clear cell component
  * Metastatic (stage IV) or recurrent disease
* Prior debulking nephrectomy required

  * Disease not amenable to complete surgical resection
* Must have HLA-identical donor

  * Matched related sibling donors must have 6/6 serologic HLA A, B, and DR match with molecular confirmation at DRB1

    * A 5/6 serologic mismatch with one antigen mismatch at locus A or B (not DR) with molecular confirmation at locus A, B, and DRB1 allowed
  * Matched unrelated donors must have a minimum of 8 out of 10 molecular matches at loci A, B, C, DRB1, and DQB1
* No brain metastases

  * Negative MRI required

PATIENT CHARACTERISTICS:

Age:

* 18 to 65

Performance status:

* Karnofsky 80-100% OR
* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin less than 2 times upper limit of normal (ULN)
* ALT/AST less than 2 times ULN
* Alkaline phosphatase less than 2 times ULN
* Hepatitis A, B, and C negative

Renal:

* Creatinine clearance greater than 50 mL/min
* Calcium less than 10.5 mg/dL (bisphosphonates allowed)

Cardiovascular:

* LVEF no less than 10% below lower limit of normal

Pulmonary:

* FEV_1 and DLCO greater than 50%

Other:

* HIV negative
* No active bacterial, fungal, or viral (including cytomegalovirus) infections
* No intolerance or allergy to tacrolimus, mycophenolate mofetil, or fludarabine
* No intolerance to 200 cGy of total body irradiation
* No other serious comorbid disease, neurologic condition, or psychosocial condition that would preclude study follow-up
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception for at least 1 month before, during, and for at least 3 months after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Prior interleukin-2 allowed
* Prior interferon alfa allowed

Chemotherapy:

* Prior chemotherapy allowed
* No other concurrent chemotherapy for RCC

Endocrine therapy:

* No concurrent corticosteroids for other comorbid disease

Radiotherapy:

* No prior extensive radiotherapy to marrow microenvironment greater than 20% of total marrow mass
* No prior radiotherapy that has reached tissue tolerance for heart, lung, liver, kidney, or spinal cord

Surgery:

* See Disease Characteristics

Other:

* No other concurrent therapy for RCC
* No concurrent enrollment on another investigational protocol for treatment of RCC
* No other concurrent immunosuppressive medications
* No other concurrent investigational drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2001-06; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary R. Hudes, MD, Study Chair — Fox Chase Cancer Center